CLINICAL TRIAL: NCT04738474
Title: Assessing and Promoting Resilience in Patients With Adult Congenital Heart Disease
Acronym: PRISMACHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jill Steiner, Assistant Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00008661; K23HL151801-01A1 (NIH)
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Congenital Heart Disease
Keywords: resilience; adult congenital heart disease; stress management; advance care planning
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRISM Intervention (Experimental): Subjects in this group will receive the PRISM intervention
  Interventions: Behavioral: Promoting Resilience in Stress Management (PRISM)
- Usual Care (Placebo Comparator): Subjects in this arm will receive usual care
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Promoting Resilience in Stress Management (PRISM) — Develops personal "resilience resources" through 1:1 sessions with a PRISM coach.
  Arms: PRISM Intervention
Other: Usual Care — No additional study-specific interaction with subjects. Subjects continue to receive usual medical care.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to evaluate the feasibility and preliminary efficacy of the Promoting Resilience in Stress Management (PRISM) intervention in patients with adult congenital heart disease.

DETAILED DESCRIPTION:
After consent is obtained, eligible patients (moderate or complex ACHD, stages B, C, or D) will complete the baseline study measures assessment and be randomized to receive PRISM or usual care (anticipated n=86, 43 per group). Patients in the intervention group will participate in the six PRISM sessions over 3 months. At 3 months following enrollment, patients in both groups will again complete study measures. We will define feasibility as a) the proportion of eligible patients who enroll and b) the proportion of patients who complete the intervention among those randomized to intervention. We will define preliminary efficacy as the change in mean resilience from baseline to 3 months after randomization between those randomized to intervention and usual care. Exploratory analyses will examine PRISM's impact on patient-centered outcomes of quality of life, symptoms of anxiety and depression, and perceived competence for health care.

ELIGIBILITY:
Inclusion Criteria:

* adults with moderate or complex ACHD, stages B, C, or D as defined by the 2018 ACHD guidelines
* receive care in our health system

Exclusion Criteria:

* diagnosis of another life-limiting illness
* inability to participate in study activities independently and in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill M Steiner, MD,MS, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Steiner JM, Marshall AR, Brumback L, Zhang YC, Glenn TM, Kovacs AH, Stout KK, Longenecker CT, Yi-Frazier JP, Rosenberg AR. A Randomized Trial of a Resilience-Building Intervention in Adult Outpatients With Congenital Heart Disease: Feasibility and Efficacy. JACC Adv. 2025 Oct;4(10 Pt 2):102164. doi: 10.1016/j.jacadv.2025.102164. Epub 2025 Sep 12. PMID 40945428
- [Derived] Steiner JM, Marshall AR, Kovacs AH, Engelberg RA, Brumback L, Stout KK, Longenecker CT, Yi-Frazier JP, Rosenberg AR. Rationale and design of a randomized controlled clinical trial of a resilience-building intervention in adults with congenital heart disease. Contemp Clin Trials. 2024 Oct;145:107638. doi: 10.1016/j.cct.2024.107638. Epub 2024 Jul 22. PMID 39047811

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Research Coordinator (RC) will screen electronic patient lists for ACHD outpatient clinics to identify potential study participants.
  RC will contact eligible patients (telephone and email), explain the study, and assess interest in participation using study team written and approved recruitment scripts.
  If agreeable, patients will be enrolled into the study. RC will obtain informed consent.
Pre-assignment Details: Enrolled participants will complete the baseline survey prior to randomization.
Groups:
- PRISM Intervention: Subjects in this group will receive the PRISM intervention. The intervention consists of a series of 5 standardized modules (plus one optional family meeting) delivered verbally in a 1:1 fashion via teleconference, roughly one every 2 weeks.
Period: Overall Study
Arm/Group | PRISM Intervention | Usual Care
Started | 40 | 38
Completed | 32 | 35
Not Completed | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRISM Intervention | Usual Care | Total
Number analyzed (Participants) | 40 | 38 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (11) | 40 (12) | 38 (12)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 20 | 28 | 48
  Gender: Male | 16 | 9 | 25
  Gender: Other | 4 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 23 | 30 | 53
  Asian | 5 | 4 | 9
  AIAN | 1 | 1 | 2
  Black/African/African American | 0 | 1 | 1
  Hispanic/Latino | 5 | 0 | 5
  Unknown | 6 | 2 | 8
Education [Count of Participants; unit: Participants]
  High School/GED | 5 | 10 | 15
  Graduate School | 14 | 9 | 23
  College | 2 | 7 | 9
  Unknown | 19 | 12 | 31
Employment [Count of Participants; unit: Participants]
  Employed | 30 | 26 | 56
  Out of Work | 7 | 8 | 15
  Student | 1 | 4 | 5
  Uknown | 2 | 0 | 2
Marital Status [Count of Participants; unit: Participants]
  Married | 24 | 24 | 48
  Single | 9 | 13 | 22
  Widowed | 0 | 1 | 1
  Divorced/Separated | 4 | 0 | 4
  Unknown | 3 | 0 | 3
ACHD Anatomy Severity [Count of Participants; unit: Participants]
  Moderate | 28 | 23 | 51
  Complex | 12 | 15 | 27
ACHD Physiology Severity [Count of Participants; unit: Participants] — Based on the ACHD Anatomy/Physiology classification as described in the 2018 Guidelines for the Care of Adults with Congenital Heart Disease; graded A-D where A is least severe physiologic impacts and D is worst.
  Participants
    C | 39 | 37 | 76
    D | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Enrollment
Description: The proportion of patients who enroll in the study among those eligible during the recruitment period
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | PRISM Intervention | Usual Care
Number analyzed (Participants) | 40 | 38
Participants | 40 | 38

2. Primary Outcome: Feasibility of PRISM
Description: The proportion of patients who complete the PRISM intervention among those randomized to intervention.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | PRISM Intervention | Usual Care
Number analyzed (Participants) | 40 | 38
Participants | 32 | 35

3. Secondary Outcome: Mean Resilience
Description: Mean (SD) resilience scores (as defined by mean CDRISC-10 score) were compared between treatment and control groups at the end of the 3-month study period. Significance of treatment effect was evaluated using the change in mean resilience (difference between scores at 3 months vs baseline). CDRISC-10: 10-item measurement of inherent resiliency, created based on the original 25-item tool. Questions revolve around personal problem-solving and approaches to adversity. Each item consists of a 5-point scale, scored from 0-4, with an overall range of 0-40 points. Higher scores indicate higher perceived resilience.
Time Frame: 3 months
Population: The difference between number of participants assigned versus here reflects dropout over the course of the study. Since our first intention was to describe feasibility, we used the enrolled numbers (40 and 38, respectively) in descriptive data analysis. For the resilience analysis, we analyzed only those with baseline and 3 months data (30 and 35, respectively).
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | PRISM Intervention | Usual Care
Number analyzed (Participants) | 30 | 35
Points | 30.1 (8.1) | 28.7 (5.8)

4. Other Pre Specified Outcome: Health-Related Quality of Life
Description: EuroQOL 5D-3L: 6-item measurement of health-related quality of life. The first 5 questions ask about symptoms and any health-related limitations. Each of these 5 items is scored on a 3-point scale, yielding a 5-digit number which can be indexed according to country (for the United States, values are -0.11 to 1). Higher scores indicate better quality of life.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | PRISM Intervention | Usual Care
Number analyzed (Participants) | 31 | 35
points | 0.9 (0.2) | 0.8 (0.2)

5. Other Pre Specified Outcome: Health-Related Quality of Life - VAS
Description: EuroQOL 5D-3L Visual Analog Scale (VAS). The final question in EuroQOL asks about health status on a visual analog scale, 0-100, where 100 is perfect health.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | PRISM Intervention | Usual Care
Number analyzed (Participants) | 31 | 35
points | 59 (14) | 73 (14)

6. Other Pre Specified Outcome: Quality of Life - LAS
Description: Single-item assessment of quality of life, continuous 0-100 scale where 100 indicates perfect quality of life.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | PRISM Intervention | Usual Care
Number analyzed (Participants) | 31 | 31
Points | 83 (12) | 79 (11)

7. Other Pre Specified Outcome: Psychological Distress
Description: Kessler-6 Psychological Distress Scale (K-6: 6-item inventory measuring the level of global psychological distress. Symptoms are rated on a 5-point scale, scored from 0-4, with an overall range of 0 to 24 points. Higher scores reflect greater distress, with scores >6 suggesting "high" distress and scores >12 suggesting "serious" distress.)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | PRISM Intervention | Usual Care
Number analyzed (Participants) | 30 | 34
Points | 5.4 (4.7) | 5.2 (4.1)

8. Other Pre Specified Outcome: Competence in Managing Healthcare
Description: Perceived Competence Scale (PCS): 4-item tool that asks about competence in managing one's disease process. Each item consists of a 7-point scale, ranging from 1 "Not at all true" to 7 "Very true." The tool is scored by calculating the mean response across all 4 questions (range 1-7). Higher scores indicate higher perceived competence.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | PRISM Intervention | Usual Care
Number analyzed (Participants) | 31 | 35
Points | 5.0 (0.9) | 5.0 (1.1)

9. Other Pre Specified Outcome: Comfort With Advance Care Planning, With Family
Time Frame: 3 months
Measure: Number; unit: Proportion of participants
Arm/Group | PRISM Intervention | Usual Care
Number analyzed (Participants) | 31 | 35
Proportion of participants | 0.4 | 0.4

10. Other Pre Specified Outcome: Comfort With Advance Care Planning, With Doctor
Time Frame: 3 months
Measure: Number; unit: Proportion of participants
Arm/Group | PRISM Intervention | Usual Care
Number analyzed (Participants) | 31 | 35
Proportion of participants | 0.5 | 0.6

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 6 months
Arm/Group | PRISM Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/38
Other Adverse Events (participants affected / at risk) | 0/40 | 0/38

LIMITATIONS AND CAVEATS:
* Dingle-site study, serving a patient population which is less racially and ethnically diverse and more highly educated than the general ACHD population.
* Decisions for a UC comparator group and to stop enrolling prior to contacting all eligible screened patients were practical decisions
* Minimally clinical important difference data is not available for these tools in ACHD
* Only evaluated intervention affect after 3 months

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT04738474/Prot_SAP_000.pdf